CLINICAL TRIAL: NCT00819962
Title: Perioperative Analgesia Using Ultrasound (US) Guided Transversus Abdominis Plane (TAP) Block
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, A.Eldawlatly, Professor of Anesthesia, King Saud University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 08-652
Record Dates: First submitted 2009-01-06; First posted 2009-01-09 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TAP (Other): ksu
  Interventions: Drug: Bupivacaine; Other: TAP

INTERVENTIONS:
Drug: Bupivacaine — Local anesthetic
Other: TAP

SUMMARY:
Perioperative analgesia using US guided TAP block

DETAILED DESCRIPTION:
Perioperative analgesia using US guided TAP block

ELIGIBILITY:
Inclusion Criteria:

* adult undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* history of cardiorespiratory disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief | after US TAP block

CONTACTS AND LOCATIONS:
Locations (1):
- A Dawlatly, Riyadh, Riyadh Region, Saudi Arabia